CLINICAL TRIAL: NCT06983717
Title: Lacrimal Deroofing for the Management of Epiphora From Lacrimal Punctal- Canalicular Abnormalities
Brief Title: Lacrimal Deroofing for Epiphora
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, Associate professor, Benha University
Other Study IDs: hamaky23
Record Dates: First submitted 2025-05-14; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Lacrimal Stenosis of Both Eyes
Keywords: lacrimal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: lacrimal deroofing — After infiltration anesthesia, patient underwent proximal lacrimal deroofing. Proper punctal dilatation is done, followed by combined 1 snip punctoplasty with a lateral canaliculotomy/ Punctotomy and posterior canaliculotomy of the lateral third. En-bloc expulsion of the concretion was done in case of canaliculitis.

SUMMARY:
Puncto-canalicular abnormalities, such as obstruction and canaliculitis, are a significant cause of epiphora. They involve proximal lacrimal drainage system. Proximal lacrimal obstructions classified into punctal stenosis canalicular obstructions. The basic principles in the treatment of punctal stenosis include creating an adequate opening, while maintaining the position of the punctum against the lacrimal lake, and preserving the lacrimal pump function. The severity of epiphora can be valued trough a grading system such as the Munk scale, fluorescein dye disappearance test, and syringing and probing and contrast dacryocystography. Canaliculitis is defined as infection of the proximal part of the lacrimal drainage system. This condition can be caused by primary infectious organisms or secondary to punctal plugs and lacrimal stents. Diagnosing canaliculitis is frequently misdiagnosed. The management includes conservative measures, local massage, syringing, and irrigation. Nevertheless, refractory cases required surgical intervention.

DETAILED DESCRIPTION:
Purpose: To report outcomes of proximal lacrimal deroofing in the management of proximal lacrimal drainage system abnormalities. Inclusion criteria: At least 18 years old patients with lacrimal punctum stenosis and/or canaliculitis. Exclusion Criteria: Trauma, Thyroid eye disease, lacrimation and other causes of epiphora. Evaluation: All patients underwent a comprehensive ophthalmic examination, and lacrimal drainage evaluation at baseline,2 weeks and 6 months after the surgery.

Outcome Measures:

Munk scale for epiphora grading (0-5); 0 No epiphora ,1 Epiphora requiring dabbing less than twice a day, 2 Epiphora requiring dabbing 2-4 times a day, 3 Epiphora requiring dabbing 5-10 times a day, 4 Epiphora requiring dabbing more than 10 times a day, 5 Constant epiphora. Grading of External Lacrimal Puncum (0-5); score 0: No papilla and punctum (punctal atresia); surgery to create a papilla, score1: Papilla is covered by a membrane; a #25 needle, followed by a punctal finder. Exudative or true membrane or fibrosis, difficult to recognize with standard punctum dilator, score 2: Less than normal size, but recognizable; a punctal finder and, then a standard punctum dilator required, score 3: Normal; regular punctum dilator required, score 4: Small slit (< 2 mm); no intervention required, score 5 Large slit (≥ 2 mm); no intervention required.

ELIGIBILITY:
Inclusion Criteria:

* epiphora due to lacrimal punctum stenosis and/or canaliculitis.

Exclusion Criteria:

• Trauma, Thyroid eye disease, lacrimation and other causes of epiphora.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: at least 18 years old patients
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Munk scale for epiphora grading (0-5) | 6 months
  0 No epiphora ,1 Epiphora requiring dabbing less than twice a day, 2 Epiphora requiring dabbing 2-4 times a day, 3 Epiphora requiring dabbing 5-10 times a day, 4 Epiphora requiring dabbing more than 10 times a day, 5 Constant epiphora.

CONTACTS AND LOCATIONS:
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
by direct contact through email
Supporting Information: Study Protocol
Time Frame: unlimited